CLINICAL TRIAL: NCT03946956
Title: Fighting Social Inequality in Cardiovascular Health I
Acronym: FISICH-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Regionshospitalet Silkeborg (Other); Vejle Hospital (Other); Svendborg Hospital (Other); Nykøbing Falster Hospital (Unknown)
Responsible Party: Principal Investigator, Jes Lindholt, Professor, Odense University Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Screening
Other Study IDs: S20160164a
Record Dates: First submitted 2019-05-09; First posted 2019-05-13 (Actual); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Cardiac Disease; Vascular Diseases
Keywords: Screening; Prevention; Cardiovascular; Public health
MeSH Terms: conditions — Heart Diseases; Vascular Diseases

STUDY DESIGN:
Intervention Model Description: 2 x factorial design regarding attendance rate to cardiovacular screening
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Prebooking (Active Comparator): Participants randomised to this arm receives a prebooked appointment to screening
  Interventions: Behavioral: Prebooking; Behavioral: Pictured invitation
- Web based booking (Placebo Comparator): Participants randomised to this arm receives an invitation to book a screening appointment webbased or by contacting the trial office.
  Interventions: Behavioral: Prebooking; Behavioral: Pictured invitation
- Pictured invitation (Active Comparator): Participants randomised to this arm receives a pictured invitation to screening
  Interventions: Behavioral: Prebooking; Behavioral: Pictured invitation
- Texted invitation (Placebo Comparator): Participants randomised to this arm receives a classical texted invitation to screening
  Interventions: Behavioral: Prebooking; Behavioral: Pictured invitation

INTERVENTIONS:
Behavioral: Prebooking — Participants are receiving a prebooked appointment for CVD screening or being invited to book an appointment for CVD Screening
Behavioral: Pictured invitation — Participants are receiving an illustrated invitation CVD screening or a classical text-invitation to book an appointment for CVD Screening

SUMMARY:
This study attempts to reduce social inequality in cardiovascular health by performing an interventional screening trial on how best to decrease cardiovascular disease (CVD) among people with low social status

DETAILED DESCRIPTION:
Background

Although CVDs have decreased, they are still among the most predominant cause of morbidity and mortality in the western world, incl. Denmark, where about 420,000 people have recognized CVD symptoms. Due to an aging population, the decline has not reduced CVD admissions and healthcare costs.

In Denmark, the CVD related hospital admission costs are DKK 4.6 billion and the pharmaceutical cost DKK 2.4 billion. The Danish National Board of Health has reported that CVD carries the second largest socioeconomic difference in burden of disease. Unfortunately, population-based health checks and screening for risk factors has proven not efficient. Consequently, screening of asymptomatic CVD is discussed intensively. In the investigators first unique CVD screening RCT (2008-11), the VIVA trial, they randomized more than 50.000 65-74 year old men for population-based ultrasound screening for abdominal aortic aneurysm (AAA), peripheral arterial disease (PAD) and hypertension. In case of positive finding, preventive medical actions were initiated. A significant reduction in overall mortality by 7% after 5 years was observed (paper submitted). Using a non-contrast CT scan, instead of the ultrasound based screening approach, has the opportunity to identify aneurysms in the entire aortic, coronary artery calcification (CAC) and arterial fibrillation, so individualized risk assessment and initiation of preventive actions on those with sign of early asymptomatic CVD is possible. The investigators therefore initiated a second trial (DANCAVAS) in 2014 randomizing 45.000 65-74 year old men with the potential of a huge beneficial effect on health, quality of life (QoL) and survival. However, screening is impaired by lower social class, and adherence to initiated prevention could be impacted as well. Consequently, they want to conduct a third RCT (FISICH) to test a number of add-ons to screening that potentially balance the benefits across socio economic groups.

The perspective is to establish a clear decision foundation for public health care policy incl. benefits, cost effectiveness and impact on social inequality of alternative variants of population screening for CVD.

Hypotheses The primary hypothesis is that an extensive circulatory screening and intervention programme reduces social inequality in cardiovascular health and fulfills the WHO criteria for screening. However, this reduction can be even more pronounced, if factors reducing the social selection to attend screening and adherence to preventive actions initiated are identified.

Aims

The aims are to

1. Test whether prebooking and/or supplemental informative pictures of the screening session and consultation improves attendance rate in general, and particular among those with the lowest educational level, lowest income level, and psychiatric disease.
2. Investigate whether confrontation of imaging of own arterial lesions at consultation after screening and/or an e-mail 3 and 12 months after the consultation in case of positive findings improves adherence to suggested cardiovascular preventive actions, and whether it influences quality of life, in general and especially concerning those with the lowest educational level, lowest income level, and psychiatric disease.

Materials and methods

In FISICH-I 20.000 60-64 year old men are randomized to the control group, while another 5.000 are randomized to the screening and intervention program for CAC, aortic and iliac aneurysms, atrial fibrillation, PAD, hypertension, diabetes and hypercholesterolaemia. There is no exclusion criteria. The screening setup is similar to DANCAVAS:

1. A small questionnaire on life style, medical history, and the QoL a.o. will be enclosed with the invitation. Non-responders are re-invited once.
2. The participant will be informed at attendance to the screening visit, and their consent will be obtained together with the questionnaire, weight, height, and waist circumference.
3. The CT scan will cover the area from the mandibular bone distally to the proximal third of the femur. Calcium scores for the common carotids, coronary arteries, aorta, and common iliac, and femoral arteries will be calculated. The aorta are visualized, and the diameter is measured in ascending, arcus, descending and abdominal, and if possible in the iliac arteries. Further the heart rhythm during the CT scan is evaluated.
4. Bilateral blood pressure will be recorded three times after 5 minutes of supine rest, and concurrently the ankle blood pressure are measured.
5. The HbA1c and lipid parameters will be measured. Biobank blood samples are then taken, centrifuged, labelled, cooled, and stored at -80 degrees Celsius.

Follow-up visit after screening If the CAC is above the median or if an aneurism of peripheral arterial disease are detected the participant is informed of the finding and its implications at a follow-up visit. At this visit, the patient will be recommended suitable prophylactic measures, including smoking cessation, walking/exercise, a lowfat diet. Additionally to start treatment with aspirin 75 mg/day and atorvastatin 40 mg/day. If an aneurism is large the patient is referred vascular surgical assessment for the repair. Otherwise, an annual check-up of the aneurism including a CT scan will be offered. If no positive findings (CAC above the median, aneurysm or PAD) are detected, the participants will be informed of the findings by e-mail or ordinary post as preferred.

Independent of the above findings, the patients will be encouraged to see their GP for further assessment if potential undiagnosed hypertension (systolic blood pressure >160 mmHg), diabetes mellitus (HbA1c >48 mmol/mol), or significant isolated hypercholesterolemia (total-cholesterol >8.0 mmol/l) are observed, as possible continuous medical treatments will be better managed by the GPs.

The GPs will be informed by a letter of all negative and positive results and the initiated actions. Additionally in the FISICH-I trial, four further randomizations are performed. In the written invitations to the screening examination two further randomizations are performed;

* prebooking versus active booking
* +/- addition of illustrations of the examinations during the screening session.

Power calculations and Randomisations

Randomisation will be performed in SPSS by providing each individual a random number from 1-20. Those numbered +16 will be invited to participate in the screening program. Those numbered 17 and 18 will be prebooked, while those numbered 19 and 20 will have to book themselves through web-booking, email or phone.

Those with an equal number (18 and 20) will receive supplemental informative pictures of the screening session.

In case of positive finding a new random number from 1-4 is given. Those numbered 3 and 4 will be confronted with imaging of their own arterial lesions, whilst others will receive standard information. Those with an equal number (2 and 4) will receive a SMS, e-mail and phone call 3 & 12 months after the consultation. If all groups after randomisations are equally sized,- 182 will only be additionally randomized to be remembered prescription renewal after 3 and 12 months, and 182 will only have been randomized to the standard of booking (Control group for all invited). If 12 months compliance to initiated preventive medication is 66%, then with 0.05 significance level, and 80% power, the smallest difference detectable is 15%, which seems clinical relevant. However, merged analyses adjusting for the other interventions will be performed reducing the smallest detectable difference and reveal potential synergistic combinations. Similar group comparisons will be performed for all randomized interventions.

Baseline variables Age, smoking, previous or current stroke, ischemic heart disease, PAD, chronic obstructive pulmonary disease, diabetes, hypertension, use of statins, useof antithrombotics, body mass index, systolic- and diastolic blood pressure, ankle brachial index, marital status, highest educational level, personal- andin house income, psychiatric morbidity defined as any diagnosis and/or use of medications for mental illness, and QoL.

Baseline and outcome variables from national registries The CPR number assigned to Danish citizens enables individual-level linkage to multiple nation-wide healthcare and administrative registries which have proved valid.

Registry-based information on outpatient visits, hospitals admissions and procedures (The Danish National Patient Registry), relevant prescribed drugs dispensed (The Danish National Prescription Registry), socio economic status etc. (Registries at Statistics Denmark) and primary care service use (National Health Insurance Service Registry) will be obtained.

Outcomes The primary outcomes are

1. Attendance to screening
2. One-year adherence to initiated lipid-lowering and/or antithrombotic medication.

Secondary outcome is:

1. QoL,

Statistical analysis Baseline characteristics will be analysed using conventional summary statistics.

Attendance rates adjusted for invitation layout and booking-method, as well as compliance one year after initiation (def.: received a prescription 9-12 months after the consultation) adjusted for image-confrontation and post-consultation phone call are compared by logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men aged 60-64 living in the municipalities of Funen, Silkeborg, Vejle and surrounding municipailties

Exclusion Criteria:

* Men not aged 60-65
* Men not living in the mentioned municipalities
* Women

Ages: 60 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Attendance rate to screening | 6 months
  The proportion of invited attending screening

SECONDARY OUTCOMES:
Quality of Life of invitation to screening | 6 months
  Quality of life measured by EurQol 5D

CONTACTS AND LOCATIONS:
Overall Officials: Jes S Lindholt, Principal Investigator — Odense University Hospital
Locations (5):
- Denmark (5):
  - Nykøbing Falster Sygehus, Nykøbing Falster
  - Odense University Hospital, Odense
  - Region Hospital Silkeborg, Silkeborg
  - Svendborg Sygehus, Svendborg
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: No
Data will be analysed on Statistics Denmarks secured server